CLINICAL TRIAL: NCT06526325
Title: The Effect of Improved Golgi Tendon Organ Stimulation From Tendon Relaxation Techniques on Pain, Range of Motion, Functionality, Endurance and Quality of Life in Patients With Cervical Disc Herniation
Brief Title: The Effect of Tendon Release Techniques in Patients With Cervical Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Hasan Aslan, Principal Investigator, Istanbul Arel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/03
Record Dates: First submitted 2024-07-03; First posted 2024-07-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cervical Disc Herniation
Keywords: disc herniation; enhanced golgi tendon organ stimulation; pain; cervical
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of enhanced Golgi tendon organ stimulation to patients (Experimental): The effect of golgi tendon organ stimulation on the symptoms will be examined after applying the improved golgi tendon organ stimulation to patients diagnosed with cervical disc herniation and having pain, limitation of movement, spasm and tenderness in the neck region.
  Interventions: Device: Enhanced golgi tendon organ stimulation

INTERVENTIONS:
Device: Enhanced golgi tendon organ stimulation — Enhanced Golgi Tendon Organ Stimulation is a method that can be used by physiotherapists and doctors. The Golgi tendon organ is the proprioceptors located in the tendon adjacent to the myotendinous junction. It is applied using two separate heads, the stimulator and the algometer. The sternocleidomastoideus, platysma, colli longus, capitis longus, scalene, rhomboid major and minor, levator scapulae and trapezius muscles and their tendons will be vibrated with a stimulator for 30 seconds, then 0.5 kilograms of pressure will be applied with an algometer from the origin to the insertion of the muscle in the region at 0.5 centimetre intervals at an angle of 90 degrees.

SUMMARY:
The goal of this clinical trial is to investigate the effect of using enhanced golgi tendon organ stimulation on symptoms in patients with cervical disc herniation. The main question[s] it aims to answer are:

* Enhanced Golgi tendon organ stimulation is effective in reducing symptoms in patients with cervical disc herniation.
* Enhanced golgi tendon organ stimulation is not effective in reducing symptoms in patients with cervical disc herniation.

Participants will receive enhanced golgi tendon organ stimulation to the Sternocleidomastoideus, platysma, longus colli, longus capitis, scalene, rhomboid major & minor, levator scapulae and trapezius muscles for 3 weeks, 2 sessions per week for 45 minutes.

DETAILED DESCRIPTION:
Participants diagnosed with cervical disc herniation will be included. Participants will receive 6 sessions of 45 minutes each, 2 sessions per week for 3 weeks. Sternocleidomastoideus, platysma, longus colli, longus capitis, scalene muscles, rhomboid major & minor, levator scapulae and trapezius muscles and tendons of these muscles will be applied.

Two separate applications are performed with the stimulator and the algometer. After increasing the blood flow in the area for 30 seconds with the vibration of the stimulator up to the point of attachment of the tendon, a pressure of 0.5 kilograms is applied at an angle of 90 degrees at 0.5 cm intervals from the origin to the insertion of the muscle in the area with an algometer made of special steel. The aim of this treatment is to stabilise the contraction and relaxation mechanism by stimulating the Golgi tendon organ and to eliminate pain by relieving spasms.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cervical disc herniation
* Volunteering for the research

Exclusion Criteria:

* Chronic bone disease
* Have had surgery for a cervical disc herniation
* Have a structural abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08-19 (Estimated)

PRIMARY OUTCOMES:
Pain assessment with algometer | baseline, immediately after the 6 weeks intervention
  The sternocleidomastoid, platysma, longus colli, longus capitis, scalene, rhomboid major and minor, levator scapulae and trapezius muscles and their tendons are compressed to 0.5 kg using an algometer. The patient's response is used to determine whether or not there is pain.
SF-36 (short form-36) | baseline, immediately after the 6 weeks intervention
  The Short Form-36 (SF-36) is a self-assessment scale and analyses 8 dimensions of health including physical function, social function, role limitations (due to physical and emotional reasons), mental health, vitality (energy), pain and general perception of health with 36 items. In scoring the scale, each sub-dimension is given a score between 0 and 100 points, where 0 points indicate that the quality of life dimension is poor and 100 points indicate that it is good.

SECONDARY OUTCOMES:
visual analogue scale (VAS) | baseline, immediately after the 6 weeks intervention
  For pain intensity according to VAS, "no pain" is usually graded as 0 points and "worst imaginable pain" as 10 points (10 cm scale). The ranges for pain intensity are <3 mild pain, 3-6 moderate pain, >6 severe pain.
assessment of joint range of motion | baseline, immediately after the 6 weeks intervention
  Range of motion of the cervical spine will be assessed with a goniometer.
Spurling Test | baseline, immediately after the 6 weeks intervention
  With the patient in an upright sitting position, the clinician flexes and laterally flexes the patient's head and applies cranial to caudal compression. The test is considered positive if there is pain, numbness and tingling. A positive spurling test indicates that there may be a problem such as a possible nerve root compression in this area. If the test is negative, it is said that nerve root compression is less likely.
Endurance Test | baseline, immediately after the 6 weeks intervention
  The patient performs flexion, extension, right lateral flexion, left lateral flexion, right rotation and left rotation. Meanwhile, the clinician maintains the position by applying the same force in the opposite direction of movement. A stopwatch is used to time the onset of pain. The longer the time, the better the outcome. A shorter time indicates a poor clinical prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: hasan aslan, Principal Investigator — AS Physiotherapy Services centre
Locations (1):
- AS Physiotherapy Services centre, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Yilmaz M, Tarakci D, Tarakci E. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation on cervical pain associated with cervical disc herniation: A randomized trial. Complement Ther Med. 2020 Mar;49:102295. doi: 10.1016/j.ctim.2019.102295. Epub 2020 Jan 3. PMID 32147037
- [Background] Yang X, Arts MP, Bartels RHMA, Vleggeert-Lankamp CLA. The type of cervical disc herniation on MRI does not correlate to clinical outcomes. Bone Joint J. 2022 Nov;104-B(11):1242-1248. doi: 10.1302/0301-620X.104B11.BJJ-2022-0657.R2. PMID 36317351